CLINICAL TRIAL: NCT00826410
Title: Prospective Study on the Value of Subcutaneous Drains in Gastrointestinal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: PD.Dr Peter Baier, university of Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 230/02
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Digestive System Diseases [C06]; Digestive System Neoplasms [C04.588.274]
Keywords: Laparotomy; Surgical site infection; Drainage
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- subcutaneous drain (Experimental): Use of subcutaneus suction drain ("Redon") after laparotomy
  Interventions: Device: Redon drain

INTERVENTIONS:
Device: Redon drain — subcutaneous suction drain after laparotomy for two days
  Other Names: subcutaneous suction drain according to Redon

SUMMARY:
The aim of the study is to determine wether subcutaneus suction drain (type redon-drain) protect against surgical side infection by laparotomy in general surgery.

DETAILED DESCRIPTION:
If subcutan drains inserted during wound closudsure after laparotomy avoid subcutaneous haematoma and seromas by suction, these drains shout protect against surgical site infections. This is the ratio why such drain are in use in many countries. To test whether this hypothesis is true or not we pland this study.

ELIGIBILITY:
Inclusion Criteria:

* indication for laparotomy
* age older 18 years
* informed consent

Exclusion Criteria:

* organ transplantation
* operation for abdominal hernia
* appendectomy by McBurney incision
* redo-operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-05; Primary Completion 2004-12 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
number of surgical site infections according to CDC guidelines after laparotomy in general surgery | 30 days after operation

SECONDARY OUTCOMES:
risk factors for surgical site infections | 30 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Peter K Baier, MD, Principal Investigator — Department of Visceral and General Surgery University of Freiburg, Germany
Locations (1):
- Department of Visceral and General Surgery , University of Freiburg, Germany, Freiburg im Breisgau, Baden-Wurttemberg, Germany